CLINICAL TRIAL: NCT00163410
Title: A Comparative Study of Inhaled Ciclesonide 200 mcg/Day vs Fluticasone Propionate 200 mcg/Day in Children With Asthma
Brief Title: Efficacy of Ciclesonide Inhaled Once Daily Versus Fluticasone Propionate Inhaled Twice Daily in Children With Asthma (4 to 15 y) (BY9010/M1-205)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-205
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Child; Fluticasone propionate; Pediatric
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to compare the efficacy of ciclesonide versus fluticasone propionate on lung function, symptoms, and use of rescue medication in children with persistent asthma. Ciclesonide will be inhaled at one dose level once daily; fluticasone propionate will be inhaled at one dose level twice daily. The study duration consists of a baseline period (2 to 4 weeks) and a treatment period (12 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* History of persistent bronchial asthma for at least 6 months
* FEV1 50-90% of predicted

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* COPD (chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* Respiratory tract infection or asthma exacerbation within the last 30 days prior to entry into the study
* History of life-threatening asthma
* Premature birth
* Current smoking
* Smoking history with either equal or more than 10 pack-years
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500
Dates: Start 2003-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
FEV1 absolute values.

SECONDARY OUTCOMES:
FEV1 as % of predicted
PEF from spirometry
diary based morning and evening PEF
diary based symptom score
diary based salbutamol MDI use
diurnal PEF fluctuation
drop-out rate due to asthma exacerbations
time until asthma exacerbation
number of symptom free- and rescue medication free days
number of days with asthma control
physical examination
vital signs
laboratory work-up
adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (10):
- India (10):
  - Altana Pharma/Nycomed, Ahmedabad
  - Altana Pharma/Nycomed, Bangalore
  - Altana Pharma/Nycomed, Chandigarh
  - Altana Pharma/Nycomed, Coimbatore
  - Altana Pharma/Nycomed, Coimbatore, Tamilnadu
  - Altana Pharma/Nycomed, Delhi
  - Altana Pharma/Nycomed, Kolkata
  - Altana Pharma/Nycomed, Mumbai
  - Altana Pharma/Nycomed, Pune
  - Altana Pharma/Nycomed, Shastri Nagar, Jaipur

REFERENCES:
- See also: BY9010_M1-205 Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4525&filename=BY9010_M1-205%20Synopsis.AZCT.com%20posting.pdf